CLINICAL TRIAL: NCT00952445
Title: A Randomized, Double-Blind, Placebo-Controlled, 4-week Study to Evaluate the Safety and Efficacy of T0903131 Besylate in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Safety and Efficacy Study of T0903131 (INT131) Besylate to Treat Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: InteKrin Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: T-131-004
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- T0903131 Besylate (Experimental): 1.0 mg
  Interventions: Drug: T0903131 Besylate
- T0903131 Besylate (higher dose) (Experimental): 10.0 mg
  Interventions: Drug: T0903131 Besylate
- Placebo (Placebo Comparator): Once daily, oral
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: T0903131 Besylate — Once daily, oral
  Other Names: INT131 Besylate
  Arms: T0903131 Besylate; T0903131 Besylate (higher dose)
Drug: Placebo — Once daily, oral
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine if repeated daily doses of T0903131 (INT131) Besylate over 4 weeks can lower fasting blood glucose in patients with Type 2 Diabetes Mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Clinical Diagnosis of Type 2 Diabetes Mellitus for at least 3 months prior to enrollment
* Fasting Plasma Glucose between 126 and 240 mg/dL
* Hemoglobin-A1c (HbA1c) between 6.8% and 10.0%
* Fasting C-peptide > 0.8 ng/mL

Exclusion Criteria:

* Treatment with any pharmacotherapy for Type 2 Diabetes Mellitus within previous 6 weeks prior to screening
* Prior treatment with Thiazolidinedione, including Troglitazone, Rosiglitazone, pioglitazone
* BMI > 42 kg/m2
* Presence of any diabetic complications requiring chronic therapy
* Presence or history of any form of hepatic disease
* Serum creatinine > 1.8 mg/dL
* History of cardiac arrhythmias or abnormal cardiac electrophysiology
* Any reason that, in the Investigator's judgment, would have interfered with the ability of the subject to comply with the requirements of the protocol

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2003-12; Study Completion 2004-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Whittier Diabetes Institute, La Jolla, California
  - Charles R. Drew University, Los Angeles, California
  - National Research Institute, Los Angeles, California
  - Lovelace Research Institute, Santa Ana, California
  - University of Miami, Miami, Florida
  - GFI Research Center, Evansville, Indiana
  - Joslin Diabetes Center, Boston, Massachusetts
  - Radiant Research, Edina, Minnesota
  - Radiant Research, St Louis, Missouri
  - St Louis Center for Clinical Research, St Louis, Missouri
  - Kaleida Health Diabetes Center, Buffalo, New York
  - Rochester Clinical Research, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Radiant Research, Portland, Oregon
  - Radiant Research, Anderson, South Carolina
  - Baylor University Endocrine Center, Dallas, Texas
  - Dallas Diabetes and Endocrine Research Center, Dallas, Texas
  - Endocrine Associates of Dallas, Dallas, Texas
  - Diabetes and Grandular Disease Clinic and Reseach Center, San Antonio, Texas
  - Endocrine Research Specialists, Ogden, Utah
  - Salem VA Medical Center, Salem, Virginia

REFERENCES:
- [Derived] Dunn FL, Higgins LS, Fredrickson J, DePaoli AM; INT131-004 study group. Selective modulation of PPARgamma activity can lower plasma glucose without typical thiazolidinedione side-effects in patients with Type 2 diabetes. J Diabetes Complications. 2011 May-Jun;25(3):151-8. doi: 10.1016/j.jdiacomp.2010.06.006. Epub 2010 Aug 23. PMID 20739195